CLINICAL TRIAL: NCT01161849
Title: Peritoneal/Serum Lactate Ratio in Relaparotomy
Brief Title: Peritoneal/ Serum Lactate Ratio in Relaparotomy
Acronym: lactate
Status: Completed | Type: Observational
Sponsor: Ospedale S. Giovanni Bosco (Other)
Responsible Party: Roberto Bini MD, Chirurgia d'urgenza
Other Study IDs: Lali2010
Record Dates: First submitted 2010-06-21; First posted 2010-07-14 (Estimated); Last update posted 2011-01-04 (Estimated); Status verified 2010-07

CONDITIONS: Surgical Complications; Relaparotomy
Keywords: lactate; urgent surgery; major surgery; surgical complications; possum; sapsII; relaparotomy

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Laparotomy performed for both emergency of elective surgery may by complicated by intrabdominal collection, anastomotic leakage, infarction and others. This conditions are able to induce peritoneal inflammation. Inflamed peritoneum are able to produce excess of lactate that the investigators can measure by collecting fluid from peritoneal drainage.

Drainage were left in abdomen for monitoring intrabdominal condition until the passage of stool or flatus. Minimum drainage of serum is present daily also in uncomplicated post operative period.

Serum lactate relates with increased systemic anaerobic metabolism such as SIRS, sepsis and systemic hypoperfusion and it is easy to measure with a blood gas analysis.

The investigators hypothesized that the increases of peritoneal/ serum lactate ratio could be an earlier, sensible, non-invasive, and economical marker of post surgical complications. The decision whether and when to perform a relaparotomy in secondary peritonitis is largely subjective and based on professional experience. Actually no existing scoring system aids in this decision.

The aim of this study is to demonstrate that this ratio could be and useful tool for the surgeon in this decisional process.

DETAILED DESCRIPTION:
Post operative intraabdominal sepsis due to surgical complications is associated with an important mortality and morbidity. Early diagnosis is crucial to improve outcome. Relaparotomy could be necessary to eradicate the intraabdominal focus of sepsis or hypoperfusion. The relaparotomy must be performed early after the diagnosis of surgical complications before the onset of multi organ failure.

This prospective observational study includes the post operative period of consecutive patients requiring both major elective surgery and urgent laparotomy.

Demographic data, presence and nature of underlying disease and surgical diagnosis will be recorded on admission and study inclusion.

Daily after study inclusion, the investigators measure: venous blood gases, blood lactate and lactate presents in the fluid collected from the abdomen. Possum and SAPSII scores will be calculated daily or when a patient develops a rapid clinical deterioration.

The investigators follow patients with complicated or uncomplicated post operative period.

Post operative complications are defined as: mesenteric ischemia, need for reintervention, anastomotic leakage or fistula, secondary peritonitis and death.

The primary end point is to demonstrate the correlation between surgical complications and serum/abdominal lactate ratio.

The second end point is to verify the correlation between need to relaparotomy and Possum an SAPSII scores.

ELIGIBILITY:
Inclusion Criteria:

* Post operative period of abdominal surgery (elective surgery of:colon-rectum, ileum, stomach and, pancreas)
* Post operative period after Urgent laparotomy for both traumatic and/or non traumatic acute abdomen
* Patients with signs of sepsis in the post operative period
* Patients with signs of systemic hypoperfusion in the post operative

Exclusion Criteria:

* Liver surgery
* Drainage of bile, blood and dejection from abdominal drainage
* Sepsis/ systemic hypoperfusion due to extraabdominal infection site

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to our surgery department for the post operative period after major abdominal surgery (neoplastic and non neoplastic) or urgent laparotomy for traumatic or non traumatic acute abdomen.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2010-08; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: roberto bini, md, Principal Investigator — Chirurgia d'urgenza; Giovanni Ferrari, MD, Principal Investigator — Medicina d'urgenza; Renzo Leli, MD, Study Chair — Chirurgia d'urgenza
Locations (2):
- Italy (2):
  - Chirurgia Generale e d'Urgenza; Ospedale SG Bosco: aslTO2, Torino, Torino
  - Medicina D'Urgenza; Ospedale SG Bosco; ASLTO2, Torino, Torino

REFERENCES:
- [Background] DeLaurier GA, Ivey RK, Johnson RH. Peritoneal fluid lactic acid and diagnostic dilemmas in acute abdominal disease. Am J Surg. 1994 Mar;167(3):302-5. doi: 10.1016/0002-9610(94)90204-6. PMID 8160901
- [Background] Paugam-Burtz C, Dupont H, Marmuse JP, Chosidow D, Malek L, Desmonts JM, Mantz J. Daily organ-system failure for diagnosis of persistent intra-abdominal sepsis after postoperative peritonitis. Intensive Care Med. 2002 May;28(5):594-8. doi: 10.1007/s00134-002-1250-5. Epub 2002 Mar 15. PMID 12029408
- [Background] Reynaert MS, Bshouty ZH, Bertrand C, Cambier-Kremer C, Calteux N, Carlier M, Col J, Tremouroux J. Early diagnosis of peritoneal infection by simultaneous measurement of lactate concentration in peritoneal fluid and blood. Intensive Care Med. 1984;10(6):301-4. doi: 10.1007/BF00254320. PMID 6512075
- [Background] van Ruler O, Lamme B, Gouma DJ, Reitsma JB, Boermeester MA. Variables associated with positive findings at relaparotomy in patients with secondary peritonitis. Crit Care Med. 2007 Feb;35(2):468-76. doi: 10.1097/01.CCM.0000253399.03545.2D. PMID 17205025
- [Background] van Ruler O, Mahler CW, Boer KR, Reuland EA, Gooszen HG, Opmeer BC, de Graaf PW, Lamme B, Gerhards MF, Steller EP, van Till JW, de Borgie CJ, Gouma DJ, Reitsma JB, Boermeester MA; Dutch Peritonitis Study Group. Comparison of on-demand vs planned relaparotomy strategy in patients with severe peritonitis: a randomized trial. JAMA. 2007 Aug 22;298(8):865-72. doi: 10.1001/jama.298.8.865. PMID 17712070
- [Background] Novotny AR, Emmanuel K, Hueser N, Knebel C, Kriner M, Ulm K, Bartels H, Siewert JR, Holzmann B. Procalcitonin ratio indicates successful surgical treatment of abdominal sepsis. Surgery. 2009 Jan;145(1):20-6. doi: 10.1016/j.surg.2008.08.009. Epub 2008 Sep 26. PMID 19081471
- [Background] Lamme B, Mahler CW, van Ruler O, Gouma DJ, Reitsma JB, Boermeester MA. Clinical predictors of ongoing infection in secondary peritonitis: systematic review. World J Surg. 2006 Dec;30(12):2170-81. doi: 10.1007/s00268-005-0333-1. PMID 17102920
- [Result] Verdant CL, Chierego M, De Moor V, Chamlou R, Creteur J, de Dieu Mutijima J, Loi P, Gelin M, Gullo A, Vincent JL, De Backer D. Prediction of postoperative complications after urgent laparotomy by intraperitoneal microdialysis: A pilot study. Ann Surg. 2006 Dec;244(6):994-1002. doi: 10.1097/01.sla.0000225092.45734.e6. PMID 17122625
- [Result] Komen N, de Bruin RW, Kleinrensink GJ, Jeekel J, Lange JF. Anastomotic leakage, the search for a reliable biomarker. A review of the literature. Colorectal Dis. 2008 Feb;10(2):109-15; discussion 115-7. doi: 10.1111/j.1463-1318.2007.01430.x. PMID 18199290
- [Derived] Bini R, Ferrari G, Apra F, Viora T, Leli R, Cotogni P. Peritoneal lactate as a potential biomarker for predicting the need for reintervention after abdominal surgery. J Trauma Acute Care Surg. 2014 Aug;77(2):376-80. doi: 10.1097/TA.0000000000000302. PMID 25058267